CLINICAL TRIAL: NCT06937619
Title: A Phase 1 Pharmacokinetic Study in Healthy Subjects to Evaluate the Relative Bioavailability of Risankizumab Following Subcutaneous Administration With On-Body Injector
Brief Title: A Study to Assess the Relative Bioavailability of Risankizumab Following Subcutaneous Administration With On-Body Injector in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M24-920
Record Dates: First submitted 2025-04-04; First posted 2025-04-22 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; Risankizumab; ABBV-066; SKYRIZI
MeSH Terms: interventions — risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Risankizumab Arm A (Experimental): Participants will receive a single dose of Risankizumab On-Body Injector (OBI) produced by new process on Day 1.
  Interventions: Drug: Risankizumab
- Risankizumab Arm B (Experimental): Participants will receive a single dose of Risankizumab On-Body Injector (OBI) produced by current process on Day 1.
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Risankizumab — Subcutaneous Injection
  Other Names: SKYRIZI; ABBV-066

SUMMARY:
This study will assess the pharmacokinetics and relative Bioavailability of risankizumab following subcutaneous (SC) administration with on-body Injector in Healthy Adult Participants.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥ 18.0 to ≤ 32.0 kg/m^2 after rounding to the tenths decimal at the time of screening. BMI is calculated as weight in kg divided by the square of height measured in meters.
* Body weight greater than 40 kg and less than 100 kg at screening.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile, and a 12-lead ECG

Exclusion Criteria:

* Previous exposure to any anti-interleukin-12/23 or anti interleukin-23 treatment for at least one year prior to Screening.
* Intention to perform strenuous exercise to which the participant is unaccustomed within one week prior to administration of first dose of study drug and during the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 263 (Actual)
Dates: Start 2025-04-21 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Risankizumab | Up to approximately 140 days
  Maximum observed plasma concentration (Cmax) of Risankizumab
Time to Cmax (Tmax) of Risankizumab | Up to approximately 140 days
  Tmax of Risankizumab
Apparent Terminal Phase Elimination Rate Constant (β) of Risankizumab | Up to approximately 140 days
  Apparent terminal phase elimination rate constant (β) of Risankizumab
Terminal Phase Elimination Half-life (t1/2) of Risankizumab | Up to approximately 140 days
  Terminal phase elimination half-life (t1/2) of Risankizumab
Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to the Last Measurable Concentration (AUCt) of Risankizumab | Up to approximately 140 days
  AUCt of Risankizumab
Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to Infinity (AUCinf) of Risankizumab | Up to approximately 140 days
  AUCinf of Risankizumab
Number of Anti-drug antibody (ADA) Titers | Up to approximately 140 days
  Incidence and concentration of anti-drug antibodies
Number of Participants Experiencing Adverse Events | Up to approximately 140 days
  An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (4):
- United States (4):
  - CenExel ACT- Anaheim Clinical Trials /ID# 274805, Anaheim, California
  - Collaborative Neuroscience Research CNS /ID# 275212, Los Alamitos, California
  - Cpmi /Id# 274464, Miami, Florida
  - Acpru /Id# 271954, Grayslake, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-920